CLINICAL TRIAL: NCT01035047
Title: Randomized Investigation of Chest Pain Diagnostic Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00010410; 1R21HL097131-01A1 (NIH)
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Acute Coronary Syndrome; Chest Pain
Keywords: Acute Coronary Syndrome; Chest pain; Cardiac MRI; Risk Stratification; Emergency Department
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Emergencies | interventions — Family Characteristics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Inpatient Care (No Intervention): This is the comparison arm. Patients are admitted to the hospital and undergo usual care.
- CDU-CMR Protocol (Experimental): Patients will be transferred to the clinical decision unit and undergo a stress cardiac MRI evaluation.
  Interventions: Other: Clinical decision unit care, coupled with cardiac MRI

INTERVENTIONS:
Other: Clinical decision unit care, coupled with cardiac MRI — After ED evaluation, patients are randomized to clinical decision unit care or inpatient care. Patients in the clinical decision unit will also undergo a stress cardiac MRI. Patients in the inpatient care arm may undergo any desired testing, including cardiac MRI, as determined by their treating physician.
  Arms: CDU-CMR Protocol

SUMMARY:
Clinical decision units (CDUs) improve resource utilization and are a recommended care option by the American College of Cardiology / American Heart Association, but are underutilized in non-low risk chest pain patients due to weaknesses of traditional cardiac testing. Cardiac magnetic resonance imaging (CMR) is sensitive and specific for ischemia, can simultaneously assess cardiac function and myocardial perfusion, and could revolutionize the diagnostic process for intermediate risk patients with chest pain. The primary objective of this trial is to measure the efficiency and safety of a combined CDU-CMR care pathway compared to inpatient care among patients with non-low risk acute chest pain.

DETAILED DESCRIPTION:
Despite spending $12 billion annually on the emergency evaluation of chest pain in the US, only 15% of admitted patients have a cardiac cause of their presenting symptoms. Clinical decision units (CDUs) improve resource utilization and are a recommended care option by the American College of Cardiology / American Heart Association, but are underutilized in non-low risk chest pain patients due to weaknesses of traditional cardiac testing. Cardiac magnetic resonance imaging (CMR) is sensitive and specific for ischemia, can simultaneously assess cardiac function and myocardial perfusion, and could revolutionize the diagnostic process for intermediate risk patients with chest pain. The superior accuracy of CMR could decrease testing and invasive procedures. The high sensitivity for ongoing ischemia could allow imaging in parallel with cardiac markers. As a result, CMR could improve the care of emergency department (ED) patients with intermediate risk chest pain. However, the efficiency and safety of CMR has not been extensively tested in the CDU setting.

Primary Hypothesis: A CDU-CMR strategy will reduce the occurrence of the composite of revascularization, re-hospitalization, and recurrent cardiac testing at 90 days when compared to an inpatient care strategy.

Methods: Participants (n=146) at intermediate risk for acute coronary syndrome (ACS) will be recruited into a clinical trial from Wake Forest University Baptist Medical Center (WFUBMC) ED. Participants will be equally randomized to CDU-CMR or inpatient care. CDU-CMR participants will undergo resting and stress CMR imaging in parallel with serial cardiac markers. Inpatient care participants will undergo serial cardiac markers followed by existing cardiac testing as determined by their care providers. The primary outcome is the composite of 90 day revascularization, re-hospitalization, and recurrent cardiac testing. The secondary outcome is index hospitalization length of stay. Safety events include ACS after discharge, mortality, and stress testing-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 21 years of age at the time of enrollment
* Chest discomfort or other symptoms consistent with possible ACS as indicated by the treating physician after obtaining an ECG and cardiac biomarkers for the patient's evaluation
* Thrombolysis in myocardial infarction (TIMI) risk score >/= 2 or physician impression of intermediate or high likelihood symptoms represent ACS
* Patient requires an inpatient or CDU evaluation for their chest pain
* The treating physician feels the patient could be discharged home if cardiac disease was excluded
* The treating physician feels the patient is safe for CDU care

Pretest probability assessment The assessment of intermediate risk for developing ACS will be based on a TIMI risk score >/= 2 and / or a board certified / board eligible emergency physician clinical impression of intermediate or high likelihood that the symptoms represent ACS. Physicians are encouraged to use the 2007 American College of Cardiology (ACC)/American Heart Association (AHA) guidelines as a framework for this assessment.

Exclusion Criteria:

* Elevated cardiac biomarkers
* New ST-segment elevation on any electrocardiogram (>/= 1 mV)
* New ST-segment depression on any electrocardiogram (>/= 2 mV)
* Known inducible cardiac ischemia without subsequent revascularization
* Unable to lie flat
* Symptomatic hypotension at the time of enrollment (systolic < 90 mm Hg)
* Contra-indications to MRI (examples: Pacemaker, defibrillator, cerebral aneurysm clips, metallic ocular foreign body, implanted devices, severe claustrophobia)
* Patient refusal or inability to comply with medical record review and follow up
* Terminal diagnosis with life expectancy less than 3 months
* Currently Pregnant
* Creatinine clearance < 45 ml/min at the time of enrollment or clinical concern for acute kidney injury
* Chronic liver disease with a creatinine clearance of <60 ml/min at the time of enrollment
* Hepato-renal syndrome
* History of liver, heart, or kidney transplant
* Confirmed angioplasty, stent placement, or coronary artery bypass grafting (CABG) within the last 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Miller, M.D., Principal Investigator — WFUBMC
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Rosamond W, Flegal K, Friday G, Furie K, Go A, Greenlund K, Haase N, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell CJ, Roger V, Rumsfeld J, Sorlie P, Steinberger J, Thom T, Wasserthiel-Smoller S, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2007 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2007 Feb 6;115(5):e69-171. doi: 10.1161/CIRCULATIONAHA.106.179918. Epub 2006 Dec 28. No abstract available. PMID 17194875
- [Background] McCaig LF, Nawar EW. National Hospital Ambulatory Medical Care Survey: 2004 emergency department summary. Adv Data. 2006 Jun 23;(372):1-29. PMID 16841785
- [Background] Christenson J, Innes G, McKnight D, Thompson CR, Wong H, Yu E, Boychuk B, Grafstein E, Rosenberg F, Gin K, Anis A, Singer J. A clinical prediction rule for early discharge of patients with chest pain. Ann Emerg Med. 2006 Jan;47(1):1-10. doi: 10.1016/j.annemergmed.2005.08.007. Epub 2005 Oct 19. PMID 16387209
- [Background] Goldstein JA, Gallagher MJ, O'Neill WW, Ross MA, O'Neil BJ, Raff GL. A randomized controlled trial of multi-slice coronary computed tomography for evaluation of acute chest pain. J Am Coll Cardiol. 2007 Feb 27;49(8):863-71. doi: 10.1016/j.jacc.2006.08.064. Epub 2007 Feb 12. PMID 17320744
- [Background] Farkouh ME, Smars PA, Reeder GS, Zinsmeister AR, Evans RW, Meloy TD, Kopecky SL, Allen M, Allison TG, Gibbons RJ, Gabriel SE. A clinical trial of a chest-pain observation unit for patients with unstable angina. Chest Pain Evaluation in the Emergency Room (CHEER) Investigators. N Engl J Med. 1998 Dec 24;339(26):1882-8. doi: 10.1056/NEJM199812243392603. PMID 9862943
- [Background] Heller GV, Stowers SA, Hendel RC, Herman SD, Daher E, Ahlberg AW, Baron JM, Mendes de Leon CF, Rizzo JA, Wackers FJ. Clinical value of acute rest technetium-99m tetrofosmin tomographic myocardial perfusion imaging in patients with acute chest pain and nondiagnostic electrocardiograms. J Am Coll Cardiol. 1998 Apr;31(5):1011-7. doi: 10.1016/s0735-1097(98)00057-6. PMID 9562001
- [Background] Sprivulis PC, Da Silva JA, Jacobs IG, Frazer AR, Jelinek GA. The association between hospital overcrowding and mortality among patients admitted via Western Australian emergency departments. Med J Aust. 2006 Mar 6;184(5):208-12. doi: 10.5694/j.1326-5377.2006.tb00416.x. PMID 16515429
- [Background] Miro O, Antonio MT, Jimenez S, De Dios A, Sanchez M, Borras A, Milla J. Decreased health care quality associated with emergency department overcrowding. Eur J Emerg Med. 1999 Jun;6(2):105-7. doi: 10.1097/00063110-199906000-00003. PMID 10461551
- [Background] Pope JH, Aufderheide TP, Ruthazer R, Woolard RH, Feldman JA, Beshansky JR, Griffith JL, Selker HP. Missed diagnoses of acute cardiac ischemia in the emergency department. N Engl J Med. 2000 Apr 20;342(16):1163-70. doi: 10.1056/NEJM200004203421603. PMID 10770981
- [Background] Braunwald E, Antman EM, Beasley JW, Califf RM, Cheitlin MD, Hochman JS, Jones RH, Kereiakes D, Kupersmith J, Levin TN, Pepine CJ, Schaeffer JW, Smith EE 3rd, Steward DE, Theroux P, Gibbons RJ, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Smith SC Jr; American College of Cardiology; American Heart Association. Committee on the Management of Patients With Unstable Angina. ACC/AHA 2002 guideline update for the management of patients with unstable angina and non-ST-segment elevation myocardial infarction--summary article: a report of the American College of Cardiology/American Heart Association task force on practice guidelines (Committee on the Management of Patients With Unstable Angina). J Am Coll Cardiol. 2002 Oct 2;40(7):1366-74. doi: 10.1016/s0735-1097(02)02336-7. No abstract available. PMID 12383588
- [Background] Hoffmann U, Nagurney JT, Moselewski F, Pena A, Ferencik M, Chae CU, Cury RC, Butler J, Abbara S, Brown DF, Manini A, Nichols JH, Achenbach S, Brady TJ. Coronary multidetector computed tomography in the assessment of patients with acute chest pain. Circulation. 2006 Nov 21;114(21):2251-60. doi: 10.1161/CIRCULATIONAHA.106.634808. Epub 2006 Oct 30. PMID 17075011
- [Background] Hollander JE, Litt HI, Chase M, Brown AM, Kim W, Baxt WG. Computed tomography coronary angiography for rapid disposition of low-risk emergency department patients with chest pain syndromes. Acad Emerg Med. 2007 Feb;14(2):112-6. doi: 10.1197/j.aem.2006.09.051. PMID 17267528
- [Background] Katz DA, Griffith JL, Beshansky JR, Selker HP. The use of empiric clinical data in the evaluation of practice guidelines for unstable angina. JAMA. 1996 Nov 20;276(19):1568-74. PMID 8918854
- [Background] Calvin JE, Klein LW, VandenBerg EJ, Meyer P, Parrillo JE. Validated risk stratification model accurately predicts low risk in patients with unstable angina. J Am Coll Cardiol. 2000 Nov 15;36(6):1803-8. doi: 10.1016/s0735-1097(00)00977-3. PMID 11092647
- [Background] Tatum JL, Jesse RL, Kontos MC, Nicholson CS, Schmidt KL, Roberts CS, Ornato JP. Comprehensive strategy for the evaluation and triage of the chest pain patient. Ann Emerg Med. 1997 Jan;29(1):116-25. doi: 10.1016/s0196-0644(97)70317-2. PMID 8998090
- [Background] Stowers SA, Eisenstein EL, Th Wackers FJ, Berman DS, Blackshear JL, Jones AD Jr, Szymanski TJ Jr, Lam LC, Simons TA, Natale D, Paige KA, Wagner GS. An economic analysis of an aggressive diagnostic strategy with single photon emission computed tomography myocardial perfusion imaging and early exercise stress testing in emergency department patients who present with chest pain but nondiagnostic electrocardiograms: results from a randomized trial. Ann Emerg Med. 2000 Jan;35(1):17-25. doi: 10.1016/S0196-0644(00)70100-4. PMID 10613936
- [Background] Gomberg-Maitland M, Murphy SA, Moliterno DJ, Cannon CP. Are we appropriately triaging patients with unstable angina? Am Heart J. 2005 Apr;149(4):613-8. doi: 10.1016/j.ahj.2004.09.035. PMID 15990742
- [Background] Committee on the Future of Emergency Care in the United States Health System. 2006. Hospital-Based Emergency Care: At the Breaking Point. Washington, DC: The National Academies Press.
- [Background] Ramakrishna G, Milavetz JJ, Zinsmeister AR, Farkouh ME, Evans RW, Allison TG, Smars PA, Gibbons RJ. Effect of exercise treadmill testing and stress imaging on the triage of patients with chest pain: CHEER substudy. Mayo Clin Proc. 2005 Mar;80(3):322-9. doi: 10.4065/80.3.322. PMID 15757012
- [Background] Gibbons RJ, Balady GJ, Bricker JT, Chaitman BR, Fletcher GF, Froelicher VF, Mark DB, McCallister BD, Mooss AN, O'Reilly MG, Winters WL, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Russell RO, Smith SC; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Committee to Update the 1997 Exercise Testing Guidelines. ACC/AHA 2002 guideline update for exercise testing: summary article. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1997 Exercise Testing Guidelines). J Am Coll Cardiol. 2002 Oct 16;40(8):1531-40. doi: 10.1016/s0735-1097(02)02164-2. No abstract available. PMID 12392846
- [Background] Detrano R, Gianrossi R, Froelicher V. The diagnostic accuracy of the exercise electrocardiogram: a meta-analysis of 22 years of research. Prog Cardiovasc Dis. 1989 Nov-Dec;32(3):173-206. doi: 10.1016/0033-0620(89)90025-x. No abstract available. PMID 2530605
- [Background] Gianrossi R, Detrano R, Mulvihill D, Lehmann K, Dubach P, Colombo A, McArthur D, Froelicher V. Exercise-induced ST depression in the diagnosis of coronary artery disease. A meta-analysis. Circulation. 1989 Jul;80(1):87-98. doi: 10.1161/01.cir.80.1.87. PMID 2661056
- [Background] Geleijnse ML, Fioretti PM, Roelandt JR. Methodology, feasibility, safety and diagnostic accuracy of dobutamine stress echocardiography. J Am Coll Cardiol. 1997 Sep;30(3):595-606. doi: 10.1016/s0735-1097(97)00206-4. PMID 9283514
- [Background] Klocke FJ, Baird MG, Lorell BH, Bateman TM, Messer JV, Berman DS, O'Gara PT, Carabello BA, Russell RO Jr, Cerqueira MD, St John Sutton MG, DeMaria AN, Udelson JE, Kennedy JW, Verani MS, Williams KA, Antman EM, Smith SC Jr, Alpert JS, Gregoratos G, Anderson JL, Hiratzka LF, Faxon DP, Hunt SA, Fuster V, Jacobs AK, Gibbons RJ, Russell RO; American College of Cardiology; American Heart Association; American Society for Nuclear Cardiology. ACC/AHA/ASNC guidelines for the clinical use of cardiac radionuclide imaging--executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (ACC/AHA/ASNC Committee to Revise the 1995 Guidelines for the Clinical Use of Cardiac Radionuclide Imaging). J Am Coll Cardiol. 2003 Oct 1;42(7):1318-33. doi: 10.1016/j.jacc.2003.08.011. No abstract available. PMID 14522503
- [Background] Hilton TC, Thompson RC, Williams HJ, Saylors R, Fulmer H, Stowers SA. Technetium-99m sestamibi myocardial perfusion imaging in the emergency room evaluation of chest pain. J Am Coll Cardiol. 1994 Apr;23(5):1016-22. doi: 10.1016/0735-1097(94)90584-3. PMID 8144763
- [Background] Kwong RY, Schussheim AE, Rekhraj S, Aletras AH, Geller N, Davis J, Christian TF, Balaban RS, Arai AE. Detecting acute coronary syndrome in the emergency department with cardiac magnetic resonance imaging. Circulation. 2003 Feb 4;107(4):531-7. doi: 10.1161/01.cir.0000047527.11221.29. PMID 12566362
- [Background] Udelson JE, Beshansky JR, Ballin DS, Feldman JA, Griffith JL, Handler J, Heller GV, Hendel RC, Pope JH, Ruthazer R, Spiegler EJ, Woolard RH, Selker HP. Myocardial perfusion imaging for evaluation and triage of patients with suspected acute cardiac ischemia: a randomized controlled trial. JAMA. 2002 Dec 4;288(21):2693-700. doi: 10.1001/jama.288.21.2693. PMID 12460092
- [Background] Manini AF, Gisondi MA, van der Vlugt TM, Schreiber DH. Adverse cardiac events in emergency department patients with chest pain six months after a negative inpatient evaluation for acute coronary syndrome. Acad Emerg Med. 2002 Sep;9(9):896-902. doi: 10.1111/j.1553-2712.2002.tb02190.x. PMID 12208678
- [Background] Desai AS, Solomon DH, Stone PH, Avorn J. Economic consequences of routine coronary angiography in low- and intermediate-risk patients with unstable angina pectoris. Am J Cardiol. 2003 Aug 15;92(4):363-7. doi: 10.1016/s0002-9149(03)00650-7. PMID 12914862
- [Background] Schneider EC, Leape LL, Weissman JS, Piana RN, Gatsonis C, Epstein AM. Racial differences in cardiac revascularization rates: does "overuse" explain higher rates among white patients? Ann Intern Med. 2001 Sep 4;135(5):328-37. doi: 10.7326/0003-4819-135-5-200109040-00009. PMID 11529696
- [Background] Cury RC, Shash K, Nagurney JT, Rosito G, Shapiro MD, Nomura CH, Abbara S, Bamberg F, Ferencik M, Schmidt EJ, Brown DF, Hoffmann U, Brady TJ. Cardiac magnetic resonance with T2-weighted imaging improves detection of patients with acute coronary syndrome in the emergency department. Circulation. 2008 Aug 19;118(8):837-44. doi: 10.1161/CIRCULATIONAHA.107.740597. Epub 2008 Aug 4. PMID 18678772
- [Background] Plein S, Greenwood JP, Ridgway JP, Cranny G, Ball SG, Sivananthan MU. Assessment of non-ST-segment elevation acute coronary syndromes with cardiac magnetic resonance imaging. J Am Coll Cardiol. 2004 Dec 7;44(11):2173-81. doi: 10.1016/j.jacc.2004.08.056. PMID 15582315
- [Background] Nagel E, Lehmkuhl HB, Bocksch W, Klein C, Vogel U, Frantz E, Ellmer A, Dreysse S, Fleck E. Noninvasive diagnosis of ischemia-induced wall motion abnormalities with the use of high-dose dobutamine stress MRI: comparison with dobutamine stress echocardiography. Circulation. 1999 Feb 16;99(6):763-70. doi: 10.1161/01.cir.99.6.763. PMID 9989961
- [Background] Hundley WG, Morgan TM, Neagle CM, Hamilton CA, Rerkpattanapipat P, Link KM. Magnetic resonance imaging determination of cardiac prognosis. Circulation. 2002 Oct 29;106(18):2328-33. doi: 10.1161/01.cir.0000036017.46437.02. PMID 12403662
- [Background] Ingkanisorn WP, Kwong RY, Bohme NS, Geller NL, Rhoads KL, Dyke CK, Paterson DI, Syed MA, Aletras AH, Arai AE. Prognosis of negative adenosine stress magnetic resonance in patients presenting to an emergency department with chest pain. J Am Coll Cardiol. 2006 Apr 4;47(7):1427-32. doi: 10.1016/j.jacc.2005.11.059. Epub 2006 Mar 20. PMID 16580532
- [Background] Patel MR, Dehmer GJ, Hirshfeld JW, Smith PK, Spertus JA; American College of Cardiology Foundation Appropriateness Criteria Task Force; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; American Association for Thoracic Surgery; American Heart Association, and the American Society of Nuclear Cardiology Endorsed by the American Society of Echocardiography; Heart Failure Society of America; Society of Cardiovascular Computed Tomography. ACCF/SCAI/STS/AATS/AHA/ASNC 2009 Appropriateness Criteria for Coronary Revascularization: a report by the American College of Cardiology Foundation Appropriateness Criteria Task Force, Society for Cardiovascular Angiography and Interventions, Society of Thoracic Surgeons, American Association for Thoracic Surgery, American Heart Association, and the American Society of Nuclear Cardiology Endorsed by the American Society of Echocardiography, the Heart Failure Society of America, and the Society of Cardiovascular Computed Tomography. J Am Coll Cardiol. 2009 Feb 10;53(6):530-53. doi: 10.1016/j.jacc.2008.10.005. PMID 19195618
- [Background] Smith SC Jr, Feldman TE, Hirshfeld JW Jr, Jacobs AK, Kern MJ, King SB 3rd, Morrison DA, O'Neill WW, Schaff HV, Whitlow PL, Williams DO, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; ACC/AHA/SCAI Writing Committee to Update the 2001 Guidelines for Percutaneous Coronary Intervention. ACC/AHA/SCAI 2005 guideline update for percutaneous coronary intervention: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (ACC/AHA/SCAI Writing Committee to Update the 2001 Guidelines for Percutaneous Coronary Intervention). J Am Coll Cardiol. 2006 Jan 3;47(1):e1-121. doi: 10.1016/j.jacc.2005.12.001. No abstract available. PMID 16386656
- [Background] Miller CD, Lindsell CJ, Khandelwal S, Chandra A, Pollack CV, Tiffany BR, Hollander JE, Gibler WB, Hoekstra JW. Is the initial diagnostic impression of "noncardiac chest pain" adequate to exclude cardiac disease? Ann Emerg Med. 2004 Dec;44(6):565-74. doi: 10.1016/j.annemergmed.2004.03.021. PMID 15573030
- [Background] Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS, Smith SC Jr, Jacobs AK, Halperin JL, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non ST-Elevation Myocardial Infarction); American College of Emergency Physicians; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; American Association of Cardiovascular and Pulmonary Rehabilitation; Society for Academic Emergency Medicine. ACC/AHA 2007 guidelines for the management of patients with unstable angina/non ST-elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non ST-Elevation Myocardial Infarction): developed in collaboration with the American College of Emergency Physicians, the Society for Cardiovascular Angiography and Interventions, and the Society of Thoracic Surgeons: endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation and the Society for Academic Emergency Medicine. Circulation. 2007 Aug 14;116(7):e148-304. doi: 10.1161/CIRCULATIONAHA.107.181940. Epub 2007 Aug 6. No abstract available. PMID 17679616
- [Background] Miller CD, Banerjee A, Mahaffey KW, Kontos MC, Fermann G, Pollack CV Jr, Antman E, Aylward P, Goodman SG, Santos R, Ferguson JJ, Califf RM, Hoekstra JW. Treatment and outcomes of patients with evolving myocardial infarction: experiences from the SYNERGY trial. Eur Heart J. 2007 May;28(9):1079-84. doi: 10.1093/eurheartj/ehm016. Epub 2007 Apr 3. PMID 17405770
- [Background] Miller CD, Fermann GJ, Lindsell CJ, Mahaffey KW, Peacock WF, Pollack CV, Hollander JE, Diercks DB, Gibler WB, Hoekstra JW; EMCREG-International itrACS Investigators. Initial risk stratification and presenting characteristics of patients with evolving myocardial infarctions. Emerg Med J. 2008 Aug;25(8):492-7. doi: 10.1136/emj.2007.052183. PMID 18660397
- [Background] Miller C, Hwang W, Hoekstra J, Lefebvre C, Case D, Hundley WG. Randomized comparison of observation unit plus stress cardiac MRI and hospital admission. Journal of Cardiovascular Magnetic Resonance 2009;11(Suppl 1):O103.
- [Background] Boden WE, O'Rourke RA, Teo KK, Hartigan PM, Maron DJ, Kostuk WJ, Knudtson M, Dada M, Casperson P, Harris CL, Chaitman BR, Shaw L, Gosselin G, Nawaz S, Title LM, Gau G, Blaustein AS, Booth DC, Bates ER, Spertus JA, Berman DS, Mancini GB, Weintraub WS; COURAGE Trial Research Group. Optimal medical therapy with or without PCI for stable coronary disease. N Engl J Med. 2007 Apr 12;356(15):1503-16. doi: 10.1056/NEJMoa070829. Epub 2007 Mar 26. PMID 17387127
- [Background] Ferreira-Gonzalez I, Permanyer-Miralda G, Busse JW, Bryant DM, Montori VM, Alonso-Coello P, Walter SD, Guyatt GH. Methodologic discussions for using and interpreting composite endpoints are limited, but still identify major concerns. J Clin Epidemiol. 2007 Jul;60(7):651-7; discussion 658-62. doi: 10.1016/j.jclinepi.2006.10.020. Epub 2007 Feb 23. PMID 17573977
- [Background] Hollander JE, Blomkalns AL, Brogan GX, Diercks DB, Field JM, Garvey JL, Gibler WB, Henry TD, Hoekstra JW, Holroyd BR, Hong Y, Kirk JD, O'Neil BJ, Jackson RE; Multidisciplinary Standardized Reporting Criteria Task Force. Standardized reporting guidelines for studies evaluating risk stratification of ED patients with potential acute coronary syndromes. Acad Emerg Med. 2004 Dec;11(12):1331-40. doi: 10.1197/j.aem.2004.08.033. No abstract available. PMID 15576525
- [Background] Kline JA, Mitchell AM, Runyon MS, Jones AE, Webb WB. Electronic medical record review as a surrogate to telephone follow-up to establish outcome for diagnostic research studies in the emergency department. Acad Emerg Med. 2005 Nov;12(11):1127-33. doi: 10.1197/j.aem.2005.04.012. Epub 2005 Sep 15. PMID 16166598
- [Background] Tsushima Y, Aoki J, Endo K. Contribution of the diagnostic test to the physician's diagnostic thinking: new method to evaluate the effect. Acad Radiol. 2003 Jul;10(7):751-5. doi: 10.1016/s1076-6332(03)80120-4. PMID 12862284
- [Background] Puskas JD, Williams WH, Mahoney EM, Huber PR, Block PC, Duke PG, Staples JR, Glas KE, Marshall JJ, Leimbach ME, McCall SA, Petersen RJ, Bailey DE, Weintraub WS, Guyton RA. Off-pump vs conventional coronary artery bypass grafting: early and 1-year graft patency, cost, and quality-of-life outcomes: a randomized trial. JAMA. 2004 Apr 21;291(15):1841-9. doi: 10.1001/jama.291.15.1841. PMID 15100202
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- [Background] Therneau TM, Grambsch PM, Fleming TR. Martingale-based residuals for survival models 10.1093/biomet/77.1.147. Biometrika 1990;77(1):147-60.
- [Background] Myocardial infarction redefined--a consensus document of The Joint European Society of Cardiology/American College of Cardiology Committee for the redefinition of myocardial infarction. Eur Heart J. 2000 Sep;21(18):1502-13. doi: 10.1053/euhj.2000.2305. PMID 10973764
- [Background] Antman EM, Cohen M, Bernink PJ, McCabe CH, Horacek T, Papuchis G, Mautner B, Corbalan R, Radley D, Braunwald E. The TIMI risk score for unstable angina/non-ST elevation MI: A method for prognostication and therapeutic decision making. JAMA. 2000 Aug 16;284(7):835-42. doi: 10.1001/jama.284.7.835. PMID 10938172
- [Background] Mahaffey KW, Puma JA, Barbagelata NA, DiCarli MF, Leesar MA, Browne KF, Eisenberg PR, Bolli R, Casas AC, Molina-Viamonte V, Orlandi C, Blevins R, Gibbons RJ, Califf RM, Granger CB. Adenosine as an adjunct to thrombolytic therapy for acute myocardial infarction: results of a multicenter, randomized, placebo-controlled trial: the Acute Myocardial Infarction STudy of ADenosine (AMISTAD) trial. J Am Coll Cardiol. 1999 Nov 15;34(6):1711-20. doi: 10.1016/s0735-1097(99)00418-0. PMID 10577561
- [Background] Ross AM, Gibbons RJ, Stone GW, Kloner RA, Alexander RW; AMISTAD-II Investigators. A randomized, double-blinded, placebo-controlled multicenter trial of adenosine as an adjunct to reperfusion in the treatment of acute myocardial infarction (AMISTAD-II). J Am Coll Cardiol. 2005 Jun 7;45(11):1775-80. doi: 10.1016/j.jacc.2005.02.061. PMID 15936605
- [Background] Karha J, Gibson CM, Murphy SA, Dibattiste PM, Cannon CP; TIMI Study Group. Safety of stress testing during the evolution of unstable angina pectoris or non-ST-elevation myocardial infarction. Am J Cardiol. 2004 Dec 15;94(12):1537-9. doi: 10.1016/j.amjcard.2004.08.033. PMID 15589011
- [Derived] Miller CD, Case LD, Little WC, Mahler SA, Burke GL, Harper EN, Lefebvre C, Hiestand B, Hoekstra JW, Hamilton CA, Hundley WG. Stress CMR reduces revascularization, hospital readmission, and recurrent cardiac testing in intermediate-risk patients with acute chest pain. JACC Cardiovasc Imaging. 2013 Jul;6(7):785-94. doi: 10.1016/j.jcmg.2012.11.022. Epub 2013 May 8. PMID 23664718

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in the Emergency Department (ED) at Wake Forest Baptist Medical Center from March 2010 to June 2011.
Pre-assignment Details: No participants were excluded from the trial prior to treatment assignment.
Groups:
- CDU-CMR Protocol: Patients will be transferred to the clinical decision unit and undergo a stress cardiac MRI evaluation.
  Clinical decision unit care, coupled with cardiac MRI : After ED evaluation, patients are randomized to clinical decision unit care or inpatient care. Patients in the clinical decision unit will also undergo a stress cardiac MRI. Patients in the inpatient care arm may undergo any desired testing, including cardiac MRI, as determined by their treating physician.
Period: Overall Study
Arm/Group | CDU-CMR Protocol | Inpatient Care
Started | 52 | 53
Completed | 52 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CDU-CMR Protocol | Inpatient Care | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 38 | 81
  >=65 years | 9 | 15 | 24
Age, Continuous [Median (Full Range); unit: years] | 54 [35 to 91] | 59 [40 to 76] | 56 [35 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 28 | 29 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 50 | 53 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 15 | 35
  White | 30 | 38 | 68
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Composite of Revascularization, Re-hospitalization, and Recurrent Cardiac Testing Through 90 Days.
Time Frame: Index Hospitalization through 90 days
Population: Data from all participants was used in the primary outcome analysis.
Measure: Number; unit: participants
Arm/Group | CDU-CMR Protocol | Inpatient Care
Number analyzed (Participants) | 52 | 53
participants | 7 | 20

2. Secondary Outcome: Length of Stay
Time Frame: Duration of Index Hospitalization, an average of 1-2 days
Population: Data from all participants was used in outcome analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | CDU-CMR Protocol | Inpatient Care
Number analyzed (Participants) | 52 | 53
hours | 21.1 [14.8 to 25.2] | 26.3 [22.7 to 44.8]

3. Secondary Outcome: Acute Coronary Syndrome
Time Frame: Index Hospitalization discharge through 90 days
Population: Data from all participants was used in outcome analysis.
Measure: Number; unit: participants
Arm/Group | CDU-CMR Protocol | Inpatient Care
Number analyzed (Participants) | 52 | 53
participants | 0 | 3

4. Secondary Outcome: Mortality
Time Frame: Index Hospitalization through 90 days
Population: Data from all participants was used for outcome analysis.
Measure: Number; unit: participants
Arm/Group | CDU-CMR Protocol | Inpatient Care
Number analyzed (Participants) | 52 | 53
participants | 0 | 0

5. Secondary Outcome: Stress Testing-related Adverse Event
Time Frame: Index Hospitalization through 90 days
Population: Data from all participants was used for outcome analysis
Measure: Number; unit: participants
Arm/Group | CDU-CMR Protocol | Inpatient Care
Number analyzed (Participants) | 52 | 53
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 Year
Description: Participants may have experienced more than one of the same type of adverse event. Participants may be counted more than once in each adverse event group or classification.
Arm/Group | CDU-CMR Protocol | Inpatient Care
Serious Adverse Events (participants affected / at risk) | 14/52 | 15/53
Other Adverse Events (participants affected / at risk) | 18/52 | 17/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDU-CMR Protocol (N=52) | Inpatient Care (N=53)
Readmission for chest pain. (Cardiac disorders) | 8 (15) | 9 (16)
Admission for syncope. (Cardiac disorders) | 1 (1) | 1 (1)
Admission for dyspnea. (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulseless Electrical Activity (PEA) Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Admission for overdose with suicidal ideation and worsening depression (Psychiatric disorders) | 1 (1) | 0 (0)
Admission for laparoscopic radical prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Admission for abdominal pain, nausea, vomiting, and diarrhea. (Gastrointestinal disorders) | 1 (1) | 1 (1)
Admission for abdominal pain. (Gastrointestinal disorders) | 1 (2) | 0 (0)
Admission for motor vehicle collision (MVC) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Underwent cardiac magnetic resonance imaging with evolving myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Admission for atrial fibrillation. (Cardiac disorders) | 1 (1) | 0 (0)
Admission for palpitations and wide-complex tachycardia. (Cardiac disorders) | 1 (1) | 0 (0)
Admission for palpitations and atrial flutter with rapid ventricular rate. (Cardiac disorders) | 1 (1) | 0 (0)
Admission for celiac arteriogram and stenting. (Surgical and medical procedures) | 1 (1) | 0 (0)
Admission for shortness of breath, dysphagia, and chest pain. (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Admission for shortness of breath. (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Developed cerebral vascular accident (CVA) after dobutamine stress echocardiogram (Nervous system disorders) | 0 (0) | 0 (0)
Admission for pneumothorax after lung biopsy. (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung biopsy positive for small cell undifferentiated carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Admission for chemotherapy and radiation therapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Admission for cough, chest pain, and pain with swallowing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Admission for cough and shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Admission for angioedema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Admission for dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Admission for lower extremity pain and suspected septic hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Admission for severe lactic acidosis secondary to diabetic ketoacidosis (DKA) (Endocrine disorders) | 0 (0) | 1 (1)
Involuntary admission for psychiatric illness (Psychiatric disorders) | 0 (0) | 1 (2)
Admission for seizure, altered consciousness, and facial fractures. (Nervous system disorders) | 0 (0) | 1 (1)
Admission for left arm numbness and chest pressure. (Cardiac disorders) | 0 (0) | 1 (1)
Admission for symptomatic cholelithiasis and laparoscopic cholecystectomy. (Surgical and medical procedures) | 0 (0) | 1 (1)
Admission for dizziness and presyncopal episodes (Nervous system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome after discharge within 90 days of index. (Cardiac disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDU-CMR Protocol (N=52) | Inpatient Care (N=53)
ED visit for abdominal pain, constipation, and chest pain. (Gastrointestinal disorders) | 1 (1) | 0 (0)
ED visit for syncopal episode. (Nervous system disorders) | 1 (1) | 0 (0)
ED visit for drainage from navel and facial numbness (Nervous system disorders) | 1 (1) | 0 (0)
ED visit for chest pain. (Cardiac disorders) | 3 (3) | 3 (3)
ED visit for abdominal pain. (Gastrointestinal disorders) | 4 (4) | 2 (3)
Negative exercise stress echocardiogram performed (Surgical and medical procedures) | 1 (1) | 0 (0)
ED visit for urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
ED visit for urinary frequency, hyperglycemia, and polydypsia (Renal and urinary disorders) | 1 (1) | 0 (0)
ED visit for back pain and rib pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ED visit for back pain and hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ED visit for abnormal glucose, diabetes, and hypertension (Endocrine disorders) | 1 (1) | 0 (0)
ED visit for high blood pressure (General disorders) | 1 (1) | 0 (0)
Early termination of cardiac MRI due to concern for extensive coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
ED visit for lower abdominal pain and rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
ED visit for near syncope and mild dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
ED visit for palpitations (Cardiac disorders) | 1 (1) | 0 (0)
ED visit for intoxication (Social circumstances) | 1 (1) | 0 (0)
ED visit for deep facial abscess. (Infections and infestations) | 1 (1) | 0 (0)
ED visit for left knee injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ED visit for chest pain and intoxication (Cardiac disorders) | 1 (1) | 0 (0)
ED visit for headache (Nervous system disorders) | 1 (1) | 0 (0)
ED visit for dyspnea and generalized weakness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ED visit for upper extremity pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ED visit for abdominal pain, vomiting, and diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
ED visit for bartholin's gland cyst. (Infections and infestations) | 0 (0) | 1 (1)
ED visit for 5th metatarsal fracture and abrasion of the right knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ED visit for knee pain and chest pain. (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ED visit for back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left against medical advice (AMA) from the ED during index hospitalization (Investigations) | 0 (0) | 1 (1)
ED visit for vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
ED visit for dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ED visit for injury to nose and face (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ED visit for weakness and numbness (Vascular disorders) | 0 (0) | 1 (1)
ED visit for motor vehicle collision (MVC) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ED visit for lower extremity pain and trouble walking (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ED visit for depression (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes